CLINICAL TRIAL: NCT05418699
Title: Real-life Data from Diabetic Patients on Closed-loop Pumps
Acronym: BLOOM
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/P02/540
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Type I diabetic patient
  Interventions: Device: closed-loop insulin pump

INTERVENTIONS:
Device: closed-loop insulin pump — Follow up of patients with real-time closed-loop insulin delivery systems

SUMMARY:
To evaluate, in real life, the effect of closed-loop devices on the improvement of glycemic control in diabetic patients managed in the endocrinology departments of secondary care hospitals.

DETAILED DESCRIPTION:
In recent years, closed-loop insulin delivery have been developed to deliver real-time glucose-responsive insulin to people with type 1 diabetes. Their use has been validated in clinical trials, but international investigative centers participating in clinical trials are not always representative of secondary care centers, and the patients they manage are also different. The eligibility criteria for participants in clinical trials are more stringent and restrictive than those of the usual patient population of diabetes/endocrinology centers. The socio-demographic characteristics of patients in clinical trials, in particular the ratio of males to females, age or ethnicity, do not necessarily reflect those observed in patients actually using the device.

ELIGIBILITY:
Inclusion Criteria:

* type I diabetic
* with a closed-loop insulin pump

Exclusion Criteria:

* under legal protection order
* patient or legal guardian objecting to the use of the data in the research

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type I diabetic patients with a closed-loop insulin pump between April 2020 and August 2023
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c level | At 3 months
  Hemoglobin A1c is an indicator of your long-term glucose levels. Normal range for the hemoglobin A1c level is between 4% and 5.6%

SECONDARY OUTCOMES:
HbA1c level | At 6 months
  Hemoglobin A1c is an indicator of your long-term glucose levels. Normal range for the hemoglobin A1c level is between 4% and 5.6%
HbA1c level | At 12 months
  Hemoglobin A1c is an indicator of your long-term glucose levels. Normal range for the hemoglobin A1c level is between 4% and 5.6%
Time in range | At 3 months
  Percentage of time spent in the target range between 70 and 180 mg/dL in the last 14 days
Time in range | At 6 months
  Percentage of time spent in the target range between 70 and 180 mg/dL in the last 14 days
Time in range | At 12 months
  Percentage of time spent in the target range between 70 and 180 mg/dL in the last 14 days
Time below range | At 3 months
  Percentage of time with glucose values below 70 mg/dL in the last 14 days
Time below range | At 6 months
  Percentage of time with glucose values below 70 mg/dL in the last 14 days
Time below range | At 12 months
  Percentage of time with glucose values below 70 mg/dL in the last 14 days
Time above range | At 3 months
  Percentage of time with glucose values above 180 mg/dL in the last 14 days
Time above range | At 6 months
  Percentage of time with glucose values above 180 mg/dL in the last 14 days
Time above range | At 12 months
  Percentage of time with glucose values above 180 mg/dL in the last 14 days
Coefficient of variation | At 3 months
  Ratio of the standard deviation divided by the mean glucose and multiplying by 100 (percentage)
Coefficient of variation | At 6 months
  Ratio of the standard deviation divided by the mean glucose and multiplying by 100 (percentage)
Coefficient of variation | At 12 months
  Ratio of the standard deviation divided by the mean glucose and multiplying by 100 (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Didier GOUET, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (5):
- France (5):
  - CH Béthune-Beuvry, Béthune
  - CH Boulogne-sur-Mer, Boulogne-sur-Mer
  - CH Dax, Dax
  - CHI Mont de Marsan et du Pays des Sources, Mont-de-Marsan
  - CH Périgueux, Périgueux

IPD SHARING:
Plan to Share IPD: Yes
The database will be made available on a general-purpose open repository. Medical Subject Headings (MESH) terms will be used to describe clinical data. International standard unit will be used. Keyword are type I diabetes, Insulin Infusion Systems, Patient Outcome Assessment
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available with publication. A Digital Object Identifier will be used.
Access Criteria: The only available version will be the locked database. With the exception of dates, all data will be made available. Dates will only be collected to verify the quality of the clinical trial execution. They do not add to the clinical question, and may be a means of indirectly identifying patients.